CLINICAL TRIAL: NCT03795272
Title: A Randomized Double-blind Placebo-controlled Phase II Trial of Rucaparib Maintenance Therapy for Patients With Locally Advanced Cervical Cancer.
Brief Title: Rucaparib Maintenance Therapy in Advanced Cervical Cancer
Acronym: MaRuC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Central and Eastern European Oncology Group (Other); North Eastern German Society of Gynaecological Oncology (Other); Belgian Gynaecological Oncology Group (Other); Princess Margaret Hospital, Canada (Other); PGOG (Polish Gynaecologic Oncology Group) (Unknown); GSO Global Clinical Research BV (Other); GCP-enhederne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENGOT-Cx7-NSGO/MaRuC
Record Dates: First submitted 2018-11-03; First posted 2019-01-07 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; rucaparib; maintenance therapy; placebo-controlled
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — rucaparib

STUDY DESIGN:
Intervention Model Description: This is a multicentre, phase 2, double-blind, placebo-controlled trial of maintenance rucaparib to obtain evidence of clinical benefit of rucaparib in locally advanced cervical cancer.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rucaparib (Experimental): Patients will be treated with active oral drug, Rucaparib twice daily for 24 months
  Interventions: Drug: Rucaparib
- Placebo (Placebo Comparator): Patients will be treated with oral placebo twice daily for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rucaparib — 2:1 randomization to receive rucaparib/placebo twice daily for 24 month
  Other Names: active maintenance
  Arms: Rucaparib
Drug: Placebo — placebo
  Other Names: matched placebo maintenance
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of PARP inhibitor, rucaparib as maintenance therapy for locally advanced cervical cancer

DETAILED DESCRIPTION:
The use of concomitant cisplatin-based chemo-radiation for cervical cancer has improved survival of locally advanced cervical cancer patients and has become the standard of care. A meta-analysis revealed that the addition of concurrent chemotherapy to radiation increased the 5-year overall survival rate by 6% (HR 0.81: 60 vs 66%), and 5-year disease-free survival rate by 8%, though there is still considerable need for improvement as most patients who relapse are incurable. The unmet need is particularly higher in patients that are at high risk of recurrence. The main negative prognostic factors are higher FIGO stage as well as the presence of positive lymph nodes. Current studies are evaluating role of adjuvant chemotherapy following chemo-radiation in locally advanced disease and will possibly improve survival by reducing risk of distant metastases, however at the cost of excessive toxicity.

PARP inhibitors have shown considerable clinical benefit especially in platinum-sensitive relapsed ovarian cancer. Several PARP inhibitors have been evaluated in other gynaecological malignancies and three PARP inhibitors (olaparib, rucaparib & niraparib) are approved by European Medicines Agency and Food & Drug Administration for treatment or as maintenance therapy in ovarian cancer. Human papillomavirus causes oxidative stress that may result in DNA single-strand breaks. In cervical cancer PARP-1 expression/activity may be up-regulated in response to the ongoing oxidative stress (HPV and inflammation), and this may promote progression. This may create a vicious circle of inflammation, PARP activation, NAD+ consumption, adenosine triphosphate consumption, necrosis, and inflammation. PARPi may limit the role of PARP-1 in promoting inflammation and oxidative stress. There is theoretical plausibility that PARPi may have a role in the treatment of cervical carcinoma.

This phase II randomized placebo-controlled double-blind study will evaluate the efficacy and safety of rucaparib as adjuvant treatment for patients with locally advanced cervical cancer who are responding to chemo-radiation. This investigator-initiated study will be performed within the GCIG/ENGOT collaboration

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell, adenocarcinoma or adenosquamous carcinoma of the cervix.
2. Patient must have completed definitive chemoradiation and is evaluated to be in complete remission 10-12 week's post definitive treatment.
3. Initial FIGO stage IIB with positive nodes (histological verification or verified by MRI/PET-CT), FIGO stages IIIA, IIIB, IVA; or any stage with para-aortic metastases (including IB and IIA with positive aortic nodes).
4. Toxicities resulting from definitive treatment must resolve to grade ≤1 prior to randomization.
5. Patient must consent that archival tumour tissue can be collected at the time of screening and used for translational studies.
6. Patient must consent to collection of whole blood and blood plasma during the study period. These samples will be stored and later used for translational studies.
7. Patient agrees to undergo all analysis; radiological examinations according to protocol.
8. The patient agrees to complete PROs (QoL questionnaire) during study treatment.
9. Patients must give informed consent.
10. Patients must be at least 18 years of age.
11. ECOG performance status 0-1
12. Serum albumin >30g/l.
13. Adequate organ function

    * Absolute neutrophil count (ANC) ≥1,500/mcL
    * Platelets >100,000/mcL
    * Haemoglobin ≥ 9g/dl (no blood transfusions for 4 weeks prior entering the trial.)
    * Serum creatinine ≤1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥50mL/min using Cockcroft-Gault formula.
    * Total bilirubin ≤1.5x ULN.
    * Alanine aminotransferase (ALT) ≤2.5x ULN
14. Life expectancy of at least 12 weeks.
15. Women of childbearing potential must use highly effective methods of birth control for the duration of study participation and for 6 months afterwards.
16. All patients: Patients should not donate blood or blood components while participating in this study and through 90 days after receipt of the final dose of IMP. -

Exclusion Criteria:

1. Histological types other than in inclusion criteria, like sarcomas, small cell carcinoma with neuroendocrine differentiation, non-epithelial cancers.
2. Concurrent cancer therapies or cancer therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biologic or hormonal therapy) within last 4 weeks.
3. Concurrent treatment with an investigational agent or participation in another clinical trial.
4. Previous malignant disease: patients are not eligible for the study if actively being treated of invasive cancer. Patients with previous malignant disease who are relapse-free and treatment-free for more than three years may enter this study. Patients with previous history of in-situ carcinoma of cervix, or non-invasive basal cell and squamous cell skin carcinoma can enter this trial.
5. Active infections or other serious underlying significant medical illness, abnormal laboratory finding or psychiatric illness/social situation that would, in the investigator's judgment, make the patient inappropriate for this study. Known active or chronic hepatitis C and/or B infection. Has known history of tuberculosis.
6. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug.
7. Any evidence of distant metastases.
8. Significant cardiovascular diseases, including uncontrolled hypertension, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months prior to randomization, congestive heart failure >NYHA II (New York Heart Association), severe peripheral vascular disease, clinically significant pericardial effusion.
9. Pregnancy or breastfeeding. Patients with preserved reproductive capacity, unwilling to use a medically acceptable method of contraception for the duration of the trial and for 6 months afterwards.
10. Known hypersensitivity to the trial drugs, or to their excipients.
11. Persons who have been committed to an institution by official or judicial order
12. Patients with dependency on the sponsor, investigator or study site -

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival in months | 42 months
  the time from randomization until the date of the first objective radiological disease progression according to investigator assessment of RECIST v1.1 or death by any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival in Sub-Population in months | 42 months
  the time from randomization until the date of the first objective radiological disease progression according to investigator assessment of RECIST v1.1 or death by any cause, whichever occurs first for the predefined study subgroups.
Patient Reported Outcomes | 42 months
  Quality of Life Questionnaire
Overall Survival in months | 60 months
  the time from randomization until the date of death by any cause

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Region Sjælland
  - Rigshospitalet, København Ø, Region Sjælland

IPD SHARING:
Plan to Share IPD: Undecided